CLINICAL TRIAL: NCT05489198
Title: Ocular Clarity After Cataract Surgery With Two Different Phacoemulsification Systems
Brief Title: Cataract Surgery Technique and Ocular Clarity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Amphia Hospital (Other)
Responsible Party: Principal Investigator, Nic J. Reus, MD, PhD, Principal Investigator, Amphia Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1900
Record Dates: First submitted 2022-07-29; First posted 2022-08-05 (Actual); Last update posted 2022-08-05 (Actual); Status verified 2022-08

CONDITIONS: Cataract
Keywords: Straylight; Phacoemulsification; Cataract
MeSH Terms: conditions — Cataract | interventions — Cataract Extraction

STUDY DESIGN:
Intervention Model Description: Prospective, comparative, single-arm, randomised, and single-centre study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Centurion (Experimental): Cataract surgery performed with the Centurion phacoemulsification system
  Interventions: Procedure: cataract surgery with Centurion phacoemulsification system
- Quatera 700 (Experimental): Cataract surgery performed with the Quatera 700 phacoemulsification system
  Interventions: Procedure: cataract surgery with Quatera 700 phacoemulsification system

INTERVENTIONS:
Procedure: cataract surgery with Centurion phacoemulsification system — Cataract surgery performed with the Centurion phacoemulsification system
  Arms: Centurion
Procedure: cataract surgery with Quatera 700 phacoemulsification system — Cataract surgery performed with the Quatera 700 phacoemulsification system
  Arms: Quatera 700

SUMMARY:
The goal of this study is to study the restoration of quality of vision, expressed as straylight, in the immediate period after cataract surgery with two different phacoemulsification technologies.

DETAILED DESCRIPTION:
Cataract is an opacification of the lens. With cataract surgery, the lens is surgically removed after which a clear artificial intraocular lens is implanted. For patients, it is important that they regain functional vision as quickly as possible after surgery as a limited vision may increase the risk of falling and increases the dependency on other people. Surgical removal of the lens is done with a phacoemulsification system. Differences between phacoemulsification systems are the used pump type, the way the needle oscillates, and the fluid dynamics of the system. It is unknown whether any of the available systems offer an advantage on the amount of corneal oedema that develops after surgery and, therefore, results in a more rapid restoration of functional vision.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cataract in both eyes,
* Having consented to and is planned to undergo cataract surgery in both eyes,
* Planned for implantation of a non-toric monofocal intraocular lens (IOL) in both eyes,
* A targeted refractive error of emmetropia,
* Corneal astigmatism of ≤1.5 D,
* Age of at least 18 years,
* Willing and able to participate in both preoperative and postoperative examinations, and
* Agreeing to sign the informed consent form.

Exclusion Criteria:

* Insufficient understanding of the Dutch language to comply with study procedures,
* Any comorbidity (other than cataract) that may significantly affect visual function and/or increase straylight and/or prolong visual recovery after surgery, such as significant macular degeneration, significant glaucoma, significant diabetic eye disease, significant ocular surface disease, cornea dystrophy, corneal opacification, significant vitreous opacities (such as asteroid hyalosis and clinically significant floaters), and history of cerebral vascular accident,
* Subjects with a history of ocular surgery (e.g., corneal refractive surgery),
* Subjects with an increased risk of complicated cataract surgery:
* Lens subluxation or (phaco)iridodonesis,
* Cataract brunescens, cataract rubra, cataract nigrans, or posterior polar cataract, and
* History of ocular trauma,
* Unability to be (reliably) measured with the C-Quant straylight meter or Pentacam corneal topographer, and
* A calculated IOL power in any eye that prohibits implantation of the same type of IOL in both eyes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
Straylight | preoperative
  Amount of straylight measured with C-Quant, expressed as log(s)
Straylight | 1-2 hours after surgery
  Amount of straylight measured with C-Quant, expressed as log(s)
Straylight | 1 day after surgery
  Amount of straylight measured with C-Quant, expressed as log(s)
Straylight | 1 week after surgery
  Amount of straylight measured with C-Quant, expressed as log(s)
Straylight | 1 month after surgery
  Amount of straylight measured with C-Quant, expressed as log(s)

SECONDARY OUTCOMES:
Corneal densitometry | preoperative
  Corneal densitometry measured with Pentacam, expressed as percentage
Corneal densitometry | 1-2 hours after surgery
  Corneal densitometry measured with Pentacam, expressed as percentage
Corneal densitometry | 1 day after surgery
  Corneal densitometry measured with Pentacam, expressed as percentage
Corneal densitometry | 1 week after surgery
  Corneal densitometry measured with Pentacam, expressed as percentage
Corneal densitometry | 1 month after surgery
  Corneal densitometry measured with Pentacam, expressed as percentage
Amount of phaco energy used | Surgery day
  Amount of phaco energy used, expressed as Cumulative Dissipated Energy (CDE, for Alcon Centurion) or as Equivalent Phaco Time (EPT, for Zeiss Quatera 700)
Amount of balanced salt solution used | Surgery day
  Amount of balanced salt solution used, expressed in milliliters
Total surgery time | Surgery day
  Total surgery time per eye
Uncorrected Distance Visual Acuity | preoperative
  Uncorrected Distance Visual Acuity, expressed as logMAR
Uncorrected Distance Visual Acuity | 1-2 hours after surgery
  Uncorrected Distance Visual Acuity, expressed as logMAR
Uncorrected Distance Visual Acuity | 1 day after surgery
  Uncorrected Distance Visual Acuity, expressed as logMAR
Uncorrected Distance Visual Acuity | 1 week after surgery
  Uncorrected Distance Visual Acuity, expressed as logMAR
Uncorrected Distance Visual Acuity | 1 month after surgery
  Uncorrected Distance Visual Acuity, expressed as logMAR
Corrected Distance Visual Acuity | preoperative
  Corrected Distance Visual Acuity, expressed as logMAR
Corrected Distance Visual Acuity | 1 day after surgery
  Corrected Distance Visual Acuity, expressed as logMAR
Corrected Distance Visual Acuity | 1 week after surgery
  Corrected Distance Visual Acuity, expressed as logMAR
Corneal pachymetry | 1 month after surgery
  Corneal thickness measured with Pentacam, expressed as um
Corneal pachymetry | preoperative
  Corneal thickness measured with Pentacam, expressed as um
Corneal pachymetry | 1-2 hours after surgery
  Corneal thickness measured with Pentacam, expressed as um
Corneal pachymetry | 1 day after surgery
  Corneal thickness measured with Pentacam, expressed as um
Corneal pachymetry | 1 week after surgery
  Corneal thickness measured with Pentacam, expressed as um
Presence of corneal oedema | preoperative
  Presence of corneal oedema with slit lamp biomicroscopy
Presence of corneal oedema | 1-2 hours after surgery
  Presence of corneal oedema with slit lamp biomicroscopy
Presence of corneal oedema | 1 day after surgery
  Presence of corneal oedema with slit lamp biomicroscopy
Presence of corneal oedema | 1 week after surgery
  Presence of corneal oedema with slit lamp biomicroscopy
Presence of corneal oedema | 1 month after surgery
  Presence of corneal oedema with slit lamp biomicroscopy
Catquest-9SF | preoperative
  Catquest-9-Short-Form patient-reported outcome measure, expressed as Rasch score (min: -6.14, max: +5.71, lower scores mean a better result) and sum score (min: 9, max: 36, lower scores mean a better result)
Catquest-9SF | 1-2 hours after surgery
  Catquest-9-Short-Form patient-reported outcome measure, expressed as Rasch score (min: -6.14, max: +5.71, lower scores mean a better result) and sum score (min: 9, max: 36, lower scores mean a better result)
Catquest-9SF | 1 day after surgery
  Catquest-9-Short-Form patient-reported outcome measure, expressed as Rasch score (min: -6.14, max: +5.71, lower scores mean a better result) and sum score (min: 9, max: 36, lower scores mean a better result)
Catquest-9SF | 1 week after surgery
  Catquest-9-Short-Form patient-reported outcome measure, expressed as Rasch score (min: -6.14, max: +5.71, lower scores mean a better result) and sum score (min: 9, max: 36, lower scores mean a better result)
Catquest-9SF | 1 month after surgery
  Catquest-9-Short-Form patient-reported outcome measure, expressed as Rasch score (min: -6.14, max: +5.71, lower scores mean a better result) and sum score (min: 9, max: 36, lower scores mean a better result)
Patient-Perceived Satisfactory Improvement in Vision | 1-2 hours after surgery
  Degree of satisfactory improvement in vision (possible answers are: a) worse, b) unchanged, c) unsatisfactory improved, d) satisfactory improved, e) good to very good improved)
Patient-Perceived Satisfactory Improvement in Vision | 1 day after surgery
  Degree of satisfactory improvement in vision (possible answers are: a) worse, b) unchanged, c) unsatisfactory improved, d) satisfactory improved, e) good to very good improved)
Patient-Perceived Satisfactory Improvement in Vision | 1 week after surgery
  Degree of satisfactory improvement in vision (possible answers are: a) worse, b) unchanged, c) unsatisfactory improved, d) satisfactory improved, e) good to very good improved)
Patient-Perceived Satisfactory Improvement in Vision | 1 month after surgery
  Degree of satisfactory improvement in vision (possible answers are: a) worse, b) unchanged, c) unsatisfactory improved, d) satisfactory improved, e) good to very good improved)

CONTACTS AND LOCATIONS:
Overall Officials: Nic J. Reus, MD, PhD, Principal Investigator — Amphia Hospital

IPD SHARING:
Plan to Share IPD: No